CLINICAL TRIAL: NCT00980538
Title: Continued Access to Etravirine (ETR) in Treatment Experienced HIV-1 Infected Subjects
Brief Title: TMC125-TiDP35-C239 - Continued Access to Etravirine (ETR) in Treatment Experienced HIV-1 Infected Participants
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR016408; TMC125-TIDP35-C239 (Other: Janssen Research & Development, LLC); 2009-013126-16 (EudraCT Number)
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Results first posted 2021-12-21 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: HIV Infections; HIV-1
Keywords: TMC125-TiDP35-C239; TMC125-C239; TMC125; HIV; Etravirine; Intelence; IntelenceTM
MeSH Terms: conditions — HIV Infections | interventions — etravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Etravirine (Experimental): Etravirine Dosed by weight up to a maximum dose of 200 milligram (mg) bid until switched to an etravirine (ETR)-based treatment regimens (i.e. commercially available and reimbursed, or accessible through another source) or local standard of care, as appropriate.
  Interventions: Drug: Etravirine

INTERVENTIONS:
Drug: Etravirine — Participants will be dosed with etravirine by weight up to a maximum dose of 200 mg bid until switched to an etravirine-based treatment regimens (i.e. commercially available and reimbursed, or accessible through another source) or local standard of care, as appropriate.

SUMMARY:
The purpose of this study is to provide etravirine (ETR) through this trial until participants can be switched to locally available ETR-based treatment regimens (that is, commercially available and reimbursed, or accessible through another source [example, access program or government program]), or local standard of care, as appropriate.

DETAILED DESCRIPTION:
This is open label continued access trial for HIV-1 infected children/adolescents who have completed treatment in clinical (parent) trial with etravirine (ETR) sponsored by/in collaboration with Janssen Research & Development and who continue to benefit from use of ETR. At baseline visit, eligibility criteria will be checked. If eligibility criteria are met, participants will either continue on ETR dose they received in previous ETR (parent) trial or on adjusted dose if required by investigator.ETR dose adjustment will be based on weight using dosing guidelines. Assessment visits are recommended every 3 months (pediatric) and 6 months (adults). For most of participant, their next visit will be final visit with data collection. New participants entering study, will have baseline visit without data collection. Thereafter visits and assessments will be performed per local standard of care and documented in the participant's medical records only. Investigators will continue to report SAEs possibly related to ETR and pregnancies to sponsor using regular reporting. Treatment will be continued until: investigator determines that participant no longer benefits from ETR treatment (e.g based on viral load); treatment limiting toxicity; loss to follow-up; consent withdrawal; pregnancy; program termination by Sponsor; ETR-based treatment regimen becomes commercially available for participant's use, and is reimbursed, or accessed by another source (e.g access/government program) in region participant is living, or participants switched to local standard of care, as appropriate. Adult participants will receive ETR 200mg BID.Pediatric participants will receive ETR, doses as received in previous ETR(parent) trial, with weight based dose adjustment if necessary.

10 to <20kg:100mg BID (4*25mg or 1 tablet 100mg) 20 to <25kg:125mg BID (5*25mg or 1 tablet 100mg+1 tablet 25mg) 25 to <30kg:150mg BID (6*25mg or 1 tablet 100mg+2 tablets 25mg) >= 30kg:200mg BID (8*25mg or 2*100mg)

ELIGIBILITY:
Inclusion Criteria:

* Participants who meet all of the following criteria are eligible for this trial: Documented HIV-1 infection
* Male or female participants, aged 2 years and older
* Successfully completed a clinical (parent) pediatric trial with ETR sponsored by or in collaboration with Janssen Research & Development, and continues to receive benefit from the use of ETR
* Participant (where appropriate, depending on age) and their parent(s) or legal representative(s) have signed the Informed Consent Form (ICF)/Assent voluntarily
* Children will be informed about the program and asked to give assent (where appropriate, depending on age)
* Negative urine pregnancy test for females of childbearing potential

Exclusion Criteria:

* Participants meeting one or more of the following criteria cannot be selected: Any condition (including but not limited to alcohol and drug use), which in the opinion of the investigator could compromise the participant's safety or adherence to treatment with ETR
* Any active clinically significant disease (e.g., pancreatitis, cardiac dysfunction) or findings of medical history, laboratory or physical examination that, in the investigator's opinion, would compromise the participant's safety during treatment with ETR
* Previously demonstrated clinically significant allergy or hypersensitivity to ETR or to any of the excipients of ETR
* Pregnant or breastfeeding
* Non-vasectomized heterosexually active boys not using safe and effective birth control methods, or not willing to continue practicing these birth control methods, during the trial and until 30 days after the end of the trial (or after the last intake of the investigational medication)
* Girls, who are sexually active and able to become pregnant, not using safe and effective birth control methods, or not willing to continue practicing these birth control methods, during the trial and until 30 days after the end of the trial (or after the last intake of the investigational medication)

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2009-12-09 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2032-01-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Sciences Ireland UC Clinical Trial, Study Director — Janssen Sciences Ireland UC
Locations (29):
- United States (4):
  - Los Angeles, California
  - Washington D.C., District of Columbia
  - New York, New York
  - Philadelphia, Pennsylvania
- Argentina (2):
  - Buenos Aires
  - Ciudad Autonoma de Buenos Aire
- Brazil (3):
  - Belo Horizonte
  - Ribeirão Preto
  - Rio de Janeiro
- Montreal, Quebec, Canada
- France (2):
  - Lyon
  - Paris
- Panama City, Panama
- Rio Piedras, Puerto Rico
- Bucharest, Romania
- South Africa (9):
  - Bloemfontein
  - Boksburg
  - Cape Town
  - Dundee
  - Durban
  - George
  - Johannesburg
  - Newtown
  - Pretoria
- Spain (3):
  - Esplugues de Llobregat
  - Madrid
  - Seville
- Thailand (2):
  - Bangkok
  - Khon Kaen

RESULTS

PARTICIPANT FLOW:
Groups:
- Etravirine: Participants who previously received etravirine (ETR) in clinical trial with ETR (NCT00254046, NCT00255099, NCT00359021, NCT00665847, NCT01504841) sponsored by/in collaboration with Janssen Research & Development and continued to benefit from its use, in countries where ETR was not commercially available, was not reimbursed, and could not be accessed through another source, or where the participant was not eligible for ongoing trials with ETR received ETR 200 milligrams (mg) twice daily (bid) in adults. Pediatric participants received ETR doses as received in previous ETR (parent) trial, with weight based dose adjustment if necessary (ETR 100 mg bid for weight 10 to less than [<] 20 kilograms [kg]; ETR 125 mg bid for weight 20 to <25 kg; ETR 150 mg bid for weight 25 to <30 kg; and 200 mg bid for weight greater than or equal to [>=] 30 kg). Treatment continued until one of the following criteria was met: participant no longer benefited from etravirine treatment, toxicity, loss to follow up, etravirine became commercially available for participants' use.
Period: Overall Study
Arm/Group | Etravirine
Started | 180
Completed | 0
Not Completed | 180
Not completed — Lost to Follow-up | 20
Not completed — Sponsor's Decision | 4
Not completed — Participant/Legal Representative Withdrew Consent/Assent | 34
Not completed — Adverse Event/HIV-Related Event/Cutaneous Event/Rash | 12
Not completed — Switch to Commercially Available Medication | 25
Not completed — Participant Non-Compliant | 9
Not completed — Investigator no Longer Thinks Participant Benefits from the ETR Treatment | 9
Not completed — Participant Ineligible to Continue the Trial | 6
Not completed — Other | 60
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Etravirine
Number analyzed (Participants) | 180
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 71
  Between 18 and 65 years | 106
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (16.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112
  Male | 68
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 11
  BRAZIL | 8
  CANADA | 1
  FRANCE | 3
  ITALY | 6
  PANAMA | 4
  ROMANIA | 1
  SOUTH AFRICA | 122
  SPAIN | 7
  THAILAND | 12
  UNITED STATES | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With At-least One Adverse Event as a Measure of Safety Until Etravirine (ETR)-Based Treatment Regimen is Commercially Available
Description: An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Time Frame: Up to 10 years and 11 months
Population: Safety analysis set included all participants who received at least one dose of etravirine.
Measure: Count of Participants; unit: Participants
Arm/Group | Etravirine
Number analyzed (Participants) | 180
Participants | 42

ADVERSE EVENTS:
Time Frame: Up to 10 years and 11 months
Description: Safety analysis set included all participants who received at least one dose of etravirine.
Arm/Group | Etravirine
All-Cause Mortality (participants affected / at risk) | 6/180
Serious Adverse Events (participants affected / at risk) | 18/180
Other Adverse Events (participants affected / at risk) | 32/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etravirine (N=180)
Myocardial Infarction (Cardiac disorders) | 1
Accidental Death (General disorders) | 1
Death (General disorders) | 1
Chronic Tonsillitis (Infections and infestations) | 1
Disseminated Tuberculosis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Brain Herniation (Injury, poisoning and procedural complications) | 1
Head Injury (Injury, poisoning and procedural complications) | 1
Limb Injury (Injury, poisoning and procedural complications) | 1
Radius Fracture (Injury, poisoning and procedural complications) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Melanoma Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to Lymph Nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Encephalopathy (Nervous system disorders) | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1
Depression (Psychiatric disorders) | 2
Acute Kidney Injury (Renal and urinary disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
Hypovolaemic Shock (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etravirine (N=180)
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Mitral Valve Incompetence (Cardiac disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Conjunctival Haemorrhage (Eye disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Aphthous Ulcer (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Odynophagia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 2
Conjunctivitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Gastroenteritis Viral (Infections and infestations) | 1
Herpes Simplex (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lice Infestation (Infections and infestations) | 1
Lower Respiratory Tract Infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral Herpes (Infections and infestations) | 2
Otitis Media (Infections and infestations) | 2
Respiratory Tract Infection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 4
Tracheobronchitis (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 5
Vulvovaginal Candidiasis (Infections and infestations) | 2
Ligament Sprain (Injury, poisoning and procedural complications) | 1
Hepatic Enzyme Increased (Investigations) | 1
Lipase Increased (Investigations) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 2
Neuropathy Peripheral (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 4
Anxiety (Psychiatric disorders) | 1
Nephropathy (Renal and urinary disorders) | 1
Amenorrhoea (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Lipoatrophy (Skin and subcutaneous tissue disorders) | 1
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 1
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1
Prurigo (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 4
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees that before he/she publishes any results of this trial, he/she shall allow at least 45 days for the Sponsor to review the pre-publication manuscript prior to submission of the manuscript to the publisher, as specified in the Clinical Trial Agreement between Institution/Investigator and Sponsor.

DOCUMENTS (2):
  • Study Protocol (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/38/NCT00980538/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT00980538/SAP_001.pdf